CLINICAL TRIAL: NCT07246733
Title: A Randomized Controlled Study on the Effect of MRJPs on Improving Ovarian Function and Endometrial Receptivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY-2025-121
Record Dates: First submitted 2025-09-03; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Diminished Ovarian Reserve (DOR); Thin Endometrium
Keywords: Ovarian reserve; Endometrial receptivity; Major Royal Jelly Proteins（MRJPs）; Reproductive health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Oral MRJPs Candy (500 mg per tablet, containing 70% MRJPs freeze-dried powder + 20% sodium cellulose + 10% microcrystalline cellulose, with an appropriate amount of arabinose), taken twice a day, 1 tablet each time, for a total of 1 menstrual cycle
  Interventions: Dietary Supplement: Oral MRJPs Candy
- Control group (Placebo Comparator): Oral placebo candy (500 mg per tablet, containing 70% whey protein powder + 20% sodium cellulose + 10% microcrystalline cellulose, with appropriate amount of arabinose), taken twice a day, 1 tablet each time, for a total of 1 menstrual cycle in the control group.
  Interventions: Dietary Supplement: Oral placebo candy

INTERVENTIONS:
Dietary Supplement: Oral MRJPs Candy — 500 mg per tablet, containing 70% MRJPs freeze-dried powder + 20% sodium cellulose + 10% microcrystalline cellulose, with an appropriate amount of arabinose, taken twice a day, 1 tablet each time, for a total of 1 menstrual cycle in the control group.
  Arms: Experimental group
Dietary Supplement: Oral placebo candy — 500 mg per tablet, containing 70% whey protein powder + 20% sodium cellulose + 10% microcrystalline cellulose, with appropriate amount of arabinose, taken twice a day, 1 tablet each time, for a total of 1 menstrual cycle in the control group.
  Arms: Control group

SUMMARY:
This study will assess the effects of the rose tablet candies produced by MRJPs on the subjects, evaluate the role of MRJPs in the ovarian function and endometrial receptivity of women, reveal the potential application value of MRJPs in reproductive health, and determine its safety and effectiveness.

DETAILED DESCRIPTION:
Ovarian reserve function and endometrial receptivity are important components of female fertility. Ovarian function is regulated by various factors, including genetics, environment, oxidative stress, inflammatory response, and endocrine regulation. Decline in ovarian function is an important factor leading to decreased fertility and perimenopausal symptoms. Endometrial receptivity refers to the ability of the endometrium to accept embryos, that is, the ability to allow the embryo to undergo processes such as positioning, adhesion, and invasion in the uterine cavity. Endometrial receptivity is a key factor for successful embryo implantation.

Royal jelly, as a natural biological nutrient, is rich in proteins, lipids, carbohydrates, vitamins, and various bioactive components. It shows various potential health benefits in promoting growth and development, regulating immune function, and antioxidation. The main active component of royal jelly - royal jelly major protein (MRJPs), has been proven to have significant effects in cell proliferation, anti-inflammatory, antioxidant, and endocrine regulation. Studies have shown that MRJPs can significantly increase serum estradiol and progesterone levels, reduce follicle-stimulating hormone and luteinizing hormone contents, increase the expression levels of estrogen receptor genes and progesterone receptor genes, increase the average thickness of the endometrium, thereby improving ovarian function and enhancing endometrial receptivity.

The ELELADY Royal Jelly Major Protein Rose Pressed Tablet Candy (Food Production License Number:SC10644070506130) has two major patent technologies. The specific detection patent technology can quickly detect the freshness of royal jelly to ensure the quality of raw materials, and the green ultrafiltration membrane separation patent technology can obtain high-purity freeze-dried powder of royal jelly major protein and bee royal jelly small molecule active essence liquid that can be stored at room temperature.

This study intends to adopt a scientific and rigorous experimental design, through the combination of clinical trials and basic experiments, strictly following ethical principles, to ensure the rights and safety of the subjects, and at the same time, adopt scientific data management and analysis methods to ensure the reliability of the research results. The conduct of this study will help reveal the potential application value of MRJPs in reproductive health, provide scientific basis for its application in regulating ovarian function and endometrial receptivity and the prevention and treatment of related diseases, and also provide new ideas and research directions for the development and application of natural products in reproductive medicine.

ELIGIBILITY:
Inclusion Criteria:

* Fertile women, aged 20 to 45 years old, with regular and normal menstrual cycles.

Exclusion Criteria:

* ① Allergic to royal jelly or its components; ② Suffering from severe chronic diseases or endocrine system disorders; ③ Pregnant or breastfeeding; ④ Undergoing hormone replacement therapy (HRT) within the last month

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Anti-Müllerian hormone | From enrollment to the end of treatment at 1 month
  Ovarian function testing indicator

SECONDARY OUTCOMES:
Sex hormone levels | From enrollment to the end of treatment at 1 month
  Basic follicle-stimulating hormone
Endometrial receptivity | From enrollment to the end of treatment at 1 month
  Ultrasound examination during the luteal phase to assess endometrial receptivity
Sex hormone levels | From enrollment to the end of treatment at 1 month
  Basic luteinizing hormone
Sex hormone levels | From enrollment to the end of treatment at 1 month
  Basal estradiol hormone

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No